CLINICAL TRIAL: NCT07286578
Title: A Prospective, Multicenter, Randomized Controlled Trial to Investigate the Value of Coronary CT Angiography in the Understanding and Management of Coronary Calcium
Brief Title: A Prospective, Multicenter, Randomized Controlled Trial to Investigate the Value of Coronary CT Angiography in the Understanding and Management of Coronary Calcium (The Optimal Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC46-THE OPTIMAL TRIAL
Record Dates: First submitted 2025-11-28; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease
Keywords: IVUS; CT
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Ischemia; Heart Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guide calcium modification strategy (Experimental): Pre-procedural CT will be used to determine lesion characteristics.
  Interventions: Device: CT(Computed Tomography) guided Percutaneous Coronary Intervention
- IVUS-guide calcium modification strategy (Active Comparator): Pre-procedural IVUS will be used to determine lesion characteristics.
  Interventions: Device: IVUS (Intravascular Ultrasound) guided Percutaneous Coronary Intervention

INTERVENTIONS:
Device: CT(Computed Tomography) guided Percutaneous Coronary Intervention — CT will be used to determine lesion characteristics and post-procedural IVUS to confirm correct implantation of stent
  Arms: CT-guide calcium modification strategy
Device: IVUS (Intravascular Ultrasound) guided Percutaneous Coronary Intervention — IVUS will be used to determine lesion characteristics and post-procedural IVUS to confirm correct implantation of stent
  Arms: IVUS-guide calcium modification strategy

SUMMARY:
The OPTIMAL randomized clinical trial has been designed to compare two imaging strategies and to test the hypothesis that a calcium modification strategy informed by coronary CT angiography (CCTA) will improve procedural efficiency and effectiveness compared with the current standard of care (IVUS-guided PCI) while achieving similar clinical outcomes in patients with hemodynamically significant calcified coronary artery disease.

DETAILED DESCRIPTION:
The OPTIMAL Trial is a prospective, multicenter, randomized controlled study evaluating whether a coronary CT angiography (CCTA)-guided calcium modification strategy can improve the treatment of patients with hemodynamically significant, calcified coronary artery disease undergoing percutaneous coronary intervention (PCI).

Seven hundred patients with flow-limiting stenosis (FFRCT ≤0.80) and moderate-to-severe calcification on CCTA will be randomized 1:1 to either CCTA-guided or intravascular ultrasound (IVUS)-guided calcium modification. The study includes two co-primary endpoints: (1) superiority in final minimal stent area assessed by IVUS, and (2) non-inferiority in 12-month target vessel failure (cardiac death, target-vessel myocardial infarction, or ischemia-driven revascularization).

CCTA-guided strategy uses advanced calcium characterization to inform pre-procedural planning and selection of plaque modification techniques. IVUS-guided strategy follows contemporary intravascular imaging-based criteria for plaque preparation and PCI optimization.

The trial aims to determine whether leveraging non-invasive CT-based calcium assessment can enhance procedural efficiency and stent results while maintaining clinical safety comparable to IVUS-guided PCI.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age and younger than 85 years old
* Subject must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia (ischemia in the absence of chest pain or other anginal equivalents), unstable angina, or acute myocardial infarction) suitable for PCI. Patients with a clinical indication for revascularization presenting with stable coronary artery disease or stabilized acute coronary syndrome defined as follows unstable angina (Braunwald class IB, IC, IIB, IIC, IIIB, IIIC), patients with NSTEMI without high-risk features such as recurrence of chest pain, ST-segment depression>1mm in ≥6 leads plus STsegment elevation in aVR, life-threatening arrhythmias, mechanical complications of MI, resuscitated cardiac arrest, GRACE risk score>140.
* All target vessels must have reference vessel diameter (visually assessed by CCTA) ≥ 2.5 mm
* Subject must provide written informed consent before any study-related procedure

Exclusion Criteria:

* STEMI as the clinical presentation.
* Uncontrolled or recurrent ventricular tachycardia.
* Hemodynamic instability.
* Hemodialysis or peritoneal dialysis.
* Left main coronary artery stenosis > 50%
* Atrial fibrillation, flutter, or arrhythmias during CT acquisition.
* Previous PCI in the target vessel or CABG.
* BMI ≥ 40 kg/m2
* Insufficient CT quality assessed by the Core lab.
* Comorbidity with life expectancy ≤ 2 years.
* Planned major cardiac or non-cardiac surgery within 24 months after the index procedure Note: Major surgery is any invasive operative procedure in which an extensive resection is performed, e.g., a body cavity is entered, organs are removed, or normal anatomy is altered. Note: Minor surgery is an operation on the superficial structures of the body or a manipulative procedure that does not involve a serious risk. Planned minor surgery is not excluded.
* The subject has received a solid organ transplant that is functioning or is active on a waiting list for any solid organ transplants with expected transplantation within 24 months.
* The subject receives immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
* The subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy) or the chest/mediastinum.
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3.
* The subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
* The subject has a history of bleeding diathesis or coagulopathy or has had a significant gastro-intestinal or significant urinary bleed within the past six months. The subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc. The subject has a life expectancy <2 years for any non-cardiac cause.
* Subject is currently participating in another investigational drug or device clinical study.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 2 years following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
* Unable to provide written informed consent (IC).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2029-12-15 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that CT-guided calcium modification results in a superior final MSA Minimal Stent Area (MSA) - Imaging Endpoint (Superiority) | Perioperative/Periprocedural
  Final post-PCI minimal stent area per target lesion, measured by independent core laboratory using intravascular ultrasound (IVUS). Assesses whether CT-guided calcium modification results in superior stent expansion compared with IVUS-guided PCI.
Target Vessel Failure (TVF) - Clinical Endpoint (Non-Inferiority) | 12 months
  Composite of cardiac death, target-vessel myocardial infarction (TV-MI), or ischemia-driven target vessel revascularization (ID-TVR). TV-MI and ID-TVR are defined according to ARC-2 and the Fourth Universal Definition of MI.

SECONDARY OUTCOMES:
Procedural efficiency: Procedure time | During PCI
  Time from first angiogram to final angiogram
Procedural efficiency:Radiation dose-area product | During PCI
  Dose-area product (DAP) recorded during PCI.
Procedural efficiency: Contrast volume | During PCI
  Total contrast volume (mL) used during PCI.IVUS-Derived Mechanistic Endpoints (Core Lab)
Procedural Efficiency: Stent Area on Immediate Post-Stent IVUS | Perioperative/Periprocedural
  MSA prior to any final IVUS-guided optimization.
Procedural Efficiency: Final Stent Area at Original Minimal Lumen Area (MLA) | Perioperative/Periprocedural
  Stent area at the co-registered site of the baseline MLA.
Procedural Efficiency: Final Stent Area at Site of Maximum Calcium Arc | Perioperative/Periprocedural
  Stent area measured at the co-registered IVUS site with maximal calcium arc
Procedural Efficiency: Final Stent Area at Site of Maximum Calcium Density | Perioperative/Periprocedural
  Stent area measured at the co-registered CT-identified region of greatest Hounsfield Unit (HU) calcium density.
Procedural Efficiency: Relative Stent Expansion | Perioperative/Periprocedural
  Percentage expansion calculated as:
  MSA ÷ mean distal reference lumen area × 100.
Procedural Efficiency: Number of Calcium Fractures | Post-modification, pre-stent
  Fractures identified on intermediary IVUS after calcium modification.
Procedural Efficiency: Change in Plaque Attenuation | Post-modification, pre-stent
  Change in IVUS plaque characteristics following calcium modification.Angiographic Endpoints
Procedural Efficiency: Final Minimal Lumen Diameter | Perioperative/Periprocedural
  Minimum lumen diameter by quantitative coronary angiography (QCA)
Procedural Efficiency: Final Percent Diameter Stenosis | Perioperative/Periprocedural
  Percent stenosis of treated lesion after PCI, by QCA
Procedural Efficiency: Final TIMI Flow Grade | Perioperative/Periprocedural
  Target vessel flow graded 0-3 based on TIMI criteria. Thrombolysis In Myocardial Infarction (TIMI) Flow Grade is a 0-3 angiographic scale used during coronary angiography to describe how well blood is flowing through a coronary artery.TIMI 0 No perfusion, TIMI 1 Penetration without perfusion, TIMI 2 Partial perfusion TIMI 3 Complete perfusion (normal flow)
Procedural Efficiency: Angiographic Complications | Day of procedure
  According to Coronary dissection (NHLBI classification)
Procedural Efficiency: Angiographic Complications | Day of procedure
  According to Coronary perforation (Ellis classification)
Procedural Efficiency: Angiographic Complications | Day of procedure
  Slow-flow / no-reflow
Procedural Efficiency: Angiographic Complications | Day of procedure
  Side branch closure (TIMI 0-1)
Clinical & Safety Outcomes: Procedural Success | Perioperative/Periprocedural
  Final stenosis <30%, TIMI 3 flow, no angiographic complications, and no in-hospital major adverse cardiac events (MACE).
Clinical & Safety Outcomes: Periprocedural Myocardial Infarction (Type 4a MI) | Day 0-1
  Defined by ARC-2 and 4th Universal Definition of MI (troponin criteria + evidence of ischemia).
Clinical & Safety Outcomes: Stent Thrombosis | Up to 12 months
  Definite or probable stent thrombosis according to ARC-2 definitions.
Patient-Reported Outcomes: Residual Angina (SAQ-7 Angina Frequency) | 12 months
  Residual angina defined as SAQ-7 Angina Frequency score <100. Angina frequency represent how often a patient has had angina (chest pain/discomfort) over a recent recall period. Reported as a 0 to 100 scale: 100 = no angina; 0 = angina occurring very frequently
Patient-Reported Outcomes: Change in Angina (SAQ-7) | Baseline to 12 months
  Change in angina frequency domain score; positive values indicate improvement. Angina frequency represent how often a patient has had angina (chest pain/discomfort) over a recent recall period. Reported as a 0 to 100 scale: 100 = no angina; 0 = angina occurring very frequently

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - HACKENSACK MERIDIAN HEALTH, Inc, Jersey City, New Jersey
  - Columbia University Irving Medical Center/NewYork-Presbyterian Hospital, New York, New York
  - Weill Medical College of Cornell University, New York, New York
- Spain (3):
  - Hospital Universitari Vall Hebron, Barcelona
  - Hospital Universitario de Leon, León
  - Hospital Universitario La Paz, Madrid
- United Kingdom (5):
  - University Hospitals of Leicester NHS Trust, Leicester
  - St Bartholomew's Hospital (Barts Health NHS Trust), London
  - St George's University Hospitals NHS Foundations Trust, London
  - Newcastle Hospitals NHS Foundations Trust, Newcastle
  - John Radcliffe Hospital, Oxford, Oxford

REFERENCES:
- [Background] Collet C, Sonck J, Vandeloo B, Mizukami T, Roosens B, Lochy S, Argacha JF, Schoors D, Colaiori I, Di Gioia G, Kodeboina M, Suzuki H, Van 't Veer M, Bartunek J, Barbato E, Cosyns B, De Bruyne B. Measurement of Hyperemic Pullback Pressure Gradients to Characterize Patterns of Coronary Atherosclerosis. J Am Coll Cardiol. 2019 Oct 8;74(14):1772-1784. doi: 10.1016/j.jacc.2019.07.072. PMID 31582137
- [Background] Tajima A, Bouisset F, Ohashi H, Sakai K, Mizukami T, Rizzini ML, Gallo D, Chiastra C, Morbiducci U, Ali ZA, Spratt JC, Ando H, Amano T, Kitslaar P, Wilgenhof A, Sonck J, De Bruyne B, Collet C. Advanced CT Imaging for the Assessment of Calcific Coronary Artery Disease and PCI Planning. J Soc Cardiovasc Angiogr Interv. 2024 Mar 26;3(3Part B):101299. doi: 10.1016/j.jscai.2024.101299. eCollection 2024 Mar. PMID 39131223
- [Background] Monizzi G, Sonck J, Nagumo S, Buytaert D, Van Hoe L, Grancini L, Bartorelli AL, Vanhoenacker P, Simons P, Bladt O, Wyffels E, De Bruyne B, Andreini D, Collet C. Quantification of calcium burden by coronary CT angiography compared to optical coherence tomography. Int J Cardiovasc Imaging. 2020 Dec;36(12):2393-2402. doi: 10.1007/s10554-020-01839-z. Epub 2020 Nov 17. PMID 33205340
- [Background] Sonck J, Nagumo S, Norgaard BL, Otake H, Ko B, Zhang J, Mizukami T, Maeng M, Andreini D, Takahashi Y, Jensen JM, Ihdayhid A, Heggermont W, Barbato E, Mileva N, Munhoz D, Bartunek J, Updegrove A, Collinsworth A, Penicka M, Van Hoe L, Leipsic J, Koo BK, De Bruyne B, Collet C. Clinical Validation of a Virtual Planner for Coronary Interventions Based on Coronary CT Angiography. JACC Cardiovasc Imaging. 2022 Jul;15(7):1242-1255. doi: 10.1016/j.jcmg.2022.02.003. Epub 2022 Apr 13. PMID 35798401
- [Background] Collet C, Collison D, Mizukami T, McCartney P, Sonck J, Ford T, Munhoz D, Berry C, De Bruyne B, Oldroyd K. Differential Improvement in Angina and Health-Related Quality of Life After PCI in Focal and Diffuse Coronary Artery Disease. JACC Cardiovasc Interv. 2022 Dec 26;15(24):2506-2518. doi: 10.1016/j.jcin.2022.09.048. Epub 2022 Nov 30. PMID 36543445